CLINICAL TRIAL: NCT00440661
Title: Exploratory Study of Some Synovial Fluid Inflammation Mediatorsunder Diacerhein in Knee Osteoarthritis Patients. Phase IV Study.
Brief Title: Exploration of the Synovial Fluid Inflammation Mediators Under Diacerhein in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires NEGMA (Industry)
Responsible Party: Patrick Darses, Negma-Lerads
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEC/ART06572N; 109196
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2007-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, IL-1
MeSH Terms: conditions — Osteoarthritis | interventions — diacerein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Diacerhein

SUMMARY:
Some inflammation mediators, notably IL-1, are implied in the joint degeneration phenomena of osteoarthritis. The aim of this study is to confirm in vivo the favourable effect of diacerhein on IL-1 and also to appreciate its effect on other synovial inflammation mediators.

ELIGIBILITY:
Inclusion Criteria:

* Painful osteoarthritis
* Hydarthrosis (synovial effusion)

Exclusion Criteria:

* large effusion
* severe pathologies
* anti-osteoarthritic treatments

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Synovial concentration of IL-1

SECONDARY OUTCOMES:
Synovial concentration of IL-6
WOMAC

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre RAYNAULD, MD, Principal Investigator — Institut de Rhumatologie de Montreal
Locations (1):
- Rheumatologic Institut of Montreal, Montreal, Quebec, Canada